CLINICAL TRIAL: NCT01442584
Title: Transplantation of Ovarian Cortex to Restore Fertility
Acronym: ovatrspl
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: hadassah, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ovarian transplant- HMO-CTIL
Record Dates: First submitted 2011-07-13; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-07

CONDITIONS: Pregnancy
Keywords: ovary; cortex; transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- fertility restoration by transplantation (Experimental): fertility restoration by transplantation of ovarian cortex slivers that were cryopreserved prior to chemotherapy
  Interventions: Procedure: ovarian transplantation

INTERVENTIONS:
Procedure: ovarian transplantation — ovarian transplantation
  Other Names: frozen thawed ovarian cortex transplantation

SUMMARY:
Ovarian transplantation has been shown to restore fertility.

DETAILED DESCRIPTION:
The investigators transplant ovarian cortex previously collected from the patient prior to cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients who froze ovarian tissue

Exclusion Criteria:

* malignant cells in ovary

Ages: 20 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
pregnancy | 3-6 months
  we will start IVF within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Revel, MD, Study Chair — Hadassah
Locations (1):
- Hadassah, Jerusalem, Israel